CLINICAL TRIAL: NCT00458328
Title: The Effect of Z-338 in Subjects With Functional Dyspepsia, Evaluate the Function of Gastro-duodenum by Ultrasound
Brief Title: The Effect of Z-338 in Subjects With Functional Dyspepsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99010208
Record Dates: First submitted 2007-04-09; First posted 2007-04-10 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Functioanl Dyspepsia
MeSH Terms: interventions — Z 338

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Z-338

SUMMARY:
Z-338; PhaseIIb, Single-centre, Randomized, Double-blind, Placebo-controlled, Parallel group study in Subjects with Functional Dyspepsia, evaluate the motility of gastro-duodenum by ultrasound

ELIGIBILITY:
Inclusion Criteria:

* Postprandial fullness, upper abdominal bloating and/or early satiety should be at least moderate for 2 days or more at the 7 days at Visit 1.
* Upper abdominal pain, upper abdominal discomfort, postprandial fullness, upper abdominal bloating, early satiety, nausea, vomit and belching should be at least moderate for at least 2 symptoms for 2 days or more at the 7 days at Visit 1.

Exclusion Criteria:

* Subjects that heartburn should be the most bothersome symptom
* Subjects presenting with primary complaints relieved by stool movements (IBS)
* Subjects with diabetes by treatment
* Subjects that heartburn should be more than moderate

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-09 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Distal stomach square, Gastric emptying, Motility index, Duodenogastric reflux index

CONTACTS AND LOCATIONS:
Overall Officials: Ken Haruma, MD, PhD, Study Chair — Kawasaki Medical School
Locations (1):
- Kawasaki Medical School, Kurashiki, Okayama-ken, Japan